CLINICAL TRIAL: NCT04164121
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, Multiple-dose, Incremental Tolerance and Pharmacokinetics Study of Phenlarmide Tablets in Chinese Healthy Adult Volunteers
Brief Title: A Clinical Study Trial of Phenlarmide in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yiling Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FLZPD1002
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Parkinson Disease
Keywords: Tolerance; Safety; Pharmacokinetic characteristics
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- FLZ-150mg experimental (Experimental): Oral administration was conducted on an empty stomach, and the drug or placebo was administered once a day on day 1 and 150mg each time from day 8 to day 17.
  Interventions: Drug: Phenlarmide Tablets
- FLZ-150mg placebo (Placebo Comparator): Oral administration was conducted on an empty stomach, and the drug or placebo was administered once a day on day 1 and 150mg each time from day 8 to day 17.
  Interventions: Drug: Placebos
- FLZ-600mg experimental (Experimental): Oral administration was conducted on an empty stomach, and the drug or placebo was administered once a day on day 1 and 600mg each time from day 8 to day 17.
  Interventions: Drug: Phenlarmide Tablets
- FLZ-600mg placebo (Placebo Comparator): Oral administration was conducted on an empty stomach, and the drug or placebo was administered once a day on day 1 and 600mg each time from day 8 to day 17.
  Interventions: Drug: Placebos
- FLZ-900mg experimental (Experimental): Oral administration was conducted on an empty stomach, and the drug or placebo was administered once a day on day 1 and 900mg each time from day 8 to day 17.
  Interventions: Drug: Phenlarmide Tablets
- FLZ-900mg placebo (Placebo Comparator): Oral administration was conducted on an empty stomach, and the drug or placebo was administered once a day on day 1 and 900mg each time from day 8 to day 17.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Phenlarmide Tablets — Oral administration was conducted on an empty stomach, and the drug was administered once a day on day 1 and once a day from day 8 to day 17.
  Other Names: FLZ
  Arms: FLZ-150mg experimental; FLZ-600mg experimental; FLZ-900mg experimental
Drug: Placebos — Oral administration was conducted on an empty stomach, and the drug was administered once a day on day 1 and once a day from day 8 to day 17.
  Other Names: FLZ-Placebos
  Arms: FLZ-150mg placebo; FLZ-600mg placebo; FLZ-900mg placebo

SUMMARY:
1. To evaluate the tolerance and safety of FLA tablets in healthy volunteers.
2. To evaluate the pharmacokinetics of FLA tablets in healthy volunteers.
3. Provide basis for dosage setting for follow-up clinical research.

ELIGIBILITY:
Inclusion Criteria:

* 1)18-65 years old (including upper and lower limits);
* 2)Men and women are not limited;
* 3)Men weigh more than 50 kg, women weigh more than 45 kg, BMI 19-28 kg/m2 (including upper and lower limits);
* 4)Understand and sign the informed consent, understand the research process and requirements, and volunteer to participate in this study.

Exclusion Criteria:

* 1)There is a history of heart, liver, kidney, respiratory, digestive tract, nervous system, endocrine, immune or hematological diseases judged by researchers as having clinical significance;
* 2)There are abnormalities in vital signs, general physical examination, laboratory examination and ECG examination, which are judged to be of clinical significance by researchers;
* 3)Any drug was taken within two weeks before the study was administered, and the researchers believe that this condition may affect the evaluation results of the study;
* 4)There is a significant history of drug allergy or hypersensitivity in food that researchers have identified as clinically significant;
* 5)The positive results of serological tests (HBsAg, anti-HCV, anti-HIV or TP-Ab) were found at the time of screening;
* 6)One year before the study was administered, some researchers believed that alcohol or drug abuse history might affect the results of this study, or that alcohol breath test or urine drug screening test were positive during screening;
* 7)Those who had smoking history within three months before the first administration or who had positive urinary cotinine test in screening stage;
* 8)Those who participated in any clinical trial within 3 months before administration;
* 9)Those who donated blood more than 400 mL or 2 units within 3 months before administration;
* 10)Do not agree to avoid the use of tobacco, alcohol or caffeine-containing beverages within 24 hours before and during the trial, or to avoid vigorous exercise, or to avoid other factors affecting drug absorption, distribution, metabolism and excretion;
* 11)Pregnant or lactating women, or those with positive serum HCG test before administration, or those who are unable or unwilling to adopt contraceptive measures approved by the researchers during the study period and within three months after the end of the study, as directed by the researchers;
* 12)Researchers do not consider it suitable for participants in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Tolerance evaluation index | From 0 to 20 days after dosing
  maximum tolerated dose (MTD), dose limited toxicity (DLT)
Tmax | From 0 to 168 hours after the first dose
  The amount of time that a drug is present at the maximum concentration in serum.
Peak Plasma Concentration (Cmax) | From 0 to 168 hours after the first dose
  The PK parameters of the plasma sample
t1/2 | From 0 to 168 hours after the first dose
  The PK parameters of the plasma sample
Vz/F | From 0 to 168 hours after the first dose
  The PK parameters of the plasma sample
CL/F | From 0 to 168 hours after the first dose
  The PK parameters of the plasma sample
Mean residence time (MRT) parameter | From 0 to 168 hours after the first dose
  The PK parameters of the plasma sample
Kel | From 0 to 168 hours after the first dose
  The PK parameters of the plasma sample
Area under the plasma concentration versus time curve (AUC0-∞) | From 0 to 168 hours after the first dose
  The PK parameters of the plasma sample
AUC0-24 | From 0 to 168 hours after the first dose
  The PK parameters of the plasma sample
AUC0-72 | From 0 to 168 hours after the first dose
  The PK parameters of the plasma sample
AUC0-last | From 0 to 168 hours after the first dose
  The PK parameters of the plasma sample
Tmax, ss | From 0 to 72 hours after the last dose
  The PK parameters of the plasma sample
Cmax, ss | From 0 to 72 hours after the last dose
  The PK parameters of the plasma sample
Cmin, ss | From 0 to 72 hours after the last dose
  The PK parameters of the plasma sample
Cavg, ss | From 0 to 72 hours after the last dose
  The PK parameters of the plasma sample
t1/2, ss | From 0 to 72 hours after the last dose
  The PK parameters of the plasma sample
AUC0-24, ss | From 0 to 72 hours after the last dose
  The PK parameters of the plasma sample
AUC0-72, ss | From 0 to 72 hours after the last dose
  The PK parameters of the plasma sample
AUC0-∞, ss | From 0 to 72 hours after the last dose
  The PK parameters of the plasma sample
AUC0-last, ss | From 0 to 72 hours after the last dose
  The PK parameters of the plasma sample

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China